CLINICAL TRIAL: NCT02528461
Title: Measuring Inflammation Cells (CD163 and CD206) With the Purpose of Examining Reduction of Fibrosis in the Liver of Chronic Hepatitis C Patients Following Treatment With the Medication Sofosbuvir
Brief Title: Macrophage Activation Markers During Sofosbuvir-based Treatment Regimes of Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCV sCD163 Sofosbuvir
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C
Keywords: Sofosbuvir; Direct acting anti-viral treatment; liver cirrhosis
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — Galactose; Gastroscopy; Sofosbuvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sofosbuvir: All patients receiving Sofosbuvir based treatment regimes during the study period will be included in the study.
  All patients will receive all interventions (galactose elimination capacity test, gastroscopy, fibroscan), except liver biopsy which the patients may decline to participate in without affecting the participation in the rest of the study. If varices are found during the gastroscopy a liver vein catheterization will be performed.
  Interventions: Drug: Galactose; Procedure: Gastroscopy; Procedure: Liver biopsy; Procedure: Fibroscan; Procedure: Liver vein catheterization; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Galactose — A test to investigate the liver's ability to metabolize galactose to glucose by injecting galactose followed by measurements of blood glucose and the quantification of galactose in the urine.
  Other Names: GEC
Procedure: Gastroscopy
Procedure: Liver biopsy
Procedure: Fibroscan
Procedure: Liver vein catheterization
Drug: Sofosbuvir

SUMMARY:
The purpose of the study is to investigate how the liver is affected with regard to inflammation and fibrosis during Sofosbuvir based treatment regimes of chronic hepatitis C.

In order to examine how the liver heals, we want to use blood samples to check for the occurrence of special liver inflammation cells (CD163 and CD206). To assess to which extent fibrosis disappear during treatment, we want to examine the liver with FibroScan (a type of ultrasound examination) and also preferably with extraction of a small tissue sample. We want to examine how the liver function as inflammation and scar tissue decrease, especially concerning the liver's ability to produce proteins. Furthermore, we want to examine with a gastroscopy, if the circulation of blood in the liver is improved after successful treatment with the expected result that potential varicose veins in the esophagus vanish.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C and initiation of sofosbuvir-based direct-acting antiviral treatment

Exclusion Criteria:

* HIV or Hepatitis B Virus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C initiating sofosbuvir-based direct-acting antiviral treatment.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Changes in the macrophage activation markers sCD163 and sCD206 | 1 year

SECONDARY OUTCOMES:
Changes in liver fibrosis with fibroscan | 1 year
  Liver fibrosis will be determined using fibroscan, and reported as changes in the amount of fibrosis in the liver
Changes in histological liver fibrosis | 1 year
  Liver fibrosis will be also be determined on liver biopsies. Determining changes in fibrosis from baseline to after treatment.
Changes in clinical status | 1 year
  Defined by the number of patients with the occurrence of cirrhosis complications, eg. ascites, hepatic encephalopathy, variceal bleeding.
Changes in hepatic venous pressure | 1 year
  Hepatic venous pressure will be assessed with liver vein catheterization before and after treatment and the results reported as changes between baseline and after treatment.
Changes in metabolic liver function determined by the galactose elimination capacity (GEC) test | 1 year
  GEC will be applied before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark